CLINICAL TRIAL: NCT00565136
Title: Evaluation of the Outcomes of Restoring Pelvic Floor Support Using TOPAS, AMS Pelvic Floor Support System, in Women With Moderate Fecal Incontinence Symptoms
Brief Title: Evaluation of Outcomes of Restoring Pelvic Floor Support With TOPAS in Women With Moderate Fecal Incontinence Symptoms
Acronym: TOPAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WC0610
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Fecal Incontinence
Keywords: Device study; Pelvic floor weakness; Fecal incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOPAS (Experimental): TOPAS AMS Pelvic Floor Repair System
  Interventions: Device: TOPAS

INTERVENTIONS:
Device: TOPAS — A mesh sling permanently implanted to increase pelvic floor support

SUMMARY:
The study purpose is to gain experience with the TOPAS system, a minimally- invasively delivered self-fixating mesh for the treatment of pelvic floor weakness in women with symptoms of moderate fecal incontinence

DETAILED DESCRIPTION:
This is a multi-center study under a common protocol. Approximately 20-30 patients will be enrolled across 5 sites in the U.S. The study population is females at least 21 years of age who have attempted but have not been satisfied with conservative therapy for their fecal incontinence symptoms. The study follow-up is two years.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 21 years of age who have evidence of pelvic floor weakness
* Females who attempted but not been satisfied with conservative therapies such as dietary changes, dietary bulking agents, biofeedback, etc.
* Subjects, who have an external anal injury, must have some voluntary sphincter control

Exclusion Criteria:

* Subjects who are unwilling or unable to sign an Informed Consent form
* Subjects who are currently pregnant or considering future child-bearing
* Subjects who are contraindicated for surgery
* Subjects who are allergic to polypropylene mesh
* Subjects who are enrolled in a concurrent clinical trial
* Subjects with previous implantation of mesh or trauma to the pelvic area
* Subjects who engage in anal receptive intercourse
* Subjects with a significant evacuation disorder such as chronic constipation
* Subjects with Crohn's Disease, ulcerative colitis or chronic diarrhea as the primary cause for fecal incontinence
* Subjects who had a hysterectomy within 6 months prior to enrollment
* Subjects with vaginal prolapse that passes the hymen
* Subjects with complete rectal prolapse
* Subjects with a history of pelvic radiation that compromises the anal canal
* Subjects who have psychiatric disturbance or debilitation as a possible cause for fecal incontinence
* Subjects with a neurological disorder such as amyotrophic lateral sclerosis, multiple sclerosis, or brain tumor as a possible cause for fecal incontinence symptoms
* Subjects with an active pelvic infection or a recto-vaginal fistula
* Subjects who have not had a negative screening exam for colon cancer within 10 years of enrollment
* Subjects who have other inappropriate conditions as determined by the physician

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Mellgren, MD, PhD, Principal Investigator — Abbott Northwestern Medical Center
Locations (5):
- United States (5):
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Christ Hospital, Cincinnati, Ohio
  - St. Lukes Hospital, Allentown, Pennsylvania
  - Sacred Heart Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenblatt P, Schumacher J, Lucente V, McNevin S, Rafferty J, Mellgren A. A preliminary evaluation of the TOPAS system for the treatment of fecal incontinence in women. Female Pelvic Med Reconstr Surg. 2014 May-Jun;20(3):155-62. doi: 10.1097/SPV.0000000000000080. PMID 24763157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at 5 U.S. study centers (medical clinics) from September 2007 to August 2008. The maximum allowed enrollment number from one site is 12.
Pre-assignment Details: After signing informed consent and prior to implant, subjects completed a 3-week bowel diary to describe the FI episodes, Fecal Incontinence Quality of Life scale, Wexner Score, Symptom Severity Scale in Fecal Incontinence, pain intensity scale, and dynamic MRI or defecography.
Groups:
- TOPAS: TOPAS AMS Pelvic Floor Repair System
  TOPAS : A mesh sling permanently implanted to increase pelvic floor support
Period: Overall Study
Arm/Group | TOPAS
Started | 29
Completed | 26
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 20-30 subjects were targeted for enrollment. There was no sample size and power analysis performed for this study.
Arm/Group | TOPAS
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White / Caucasian | 28
  Other | 1
Height [Mean (Standard Deviation); unit: cm] | 164.8 (5.9)
Weight [Mean (Standard Deviation); unit: kg] | 76.3 (19.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/[m]^2] — Body Mass Index is calculated as by the formula: weight (kg) / [height (m)]^2
  kg/[m]^2 | 28.1 (7.1)
Gravidity [Mean (Standard Deviation); unit: pregnancies] — Gravidity is defined as the number of times a female has been pregnant.
  pregnancies | 3.6 (2.1)
Parity [Mean (Standard Deviation); unit: births] — Parity is defined as the number of times a female has given birth.
  births | 2.9 (1.1)
Number Cesarean Births [Mean (Standard Deviation); unit: deliveries] | 0.1 (0.3)
Number of Vaginal Births [Mean (Standard Deviation); unit: deliveries] | 2.8 (1.1)
Menopausal Status [Number; unit: participants]
  Pre-menopausal | 7
  Post-menopausal | 22
Fecal Incontinence Treatment History (failed modalities) [Number; unit: participants] — Participants can have multiple failed modalities
  participants
    Diet modification | 25
    FI medication | 9
    Biofeedback | 11
    Pelvic surgery | 3
    Other | 6
Etiology of Fecal Incontinence [Number; unit: participants] — Participants can have multiple etiologies
  participants
    Neurological | 2
    Anorectal trauma | 4
    Obstetric trauma | 10
    Idiopathic/Unknown | 15
    Congenital abnormality | 0
    Other | 0
Colonoscopy within past 10 years [Number; unit: participants]
  Yes | 24
  No | 5
Colonoscopy Results [Number; unit: participants]
  Normal | 15
  Abnormal | 8
  Unknown | 6
  Other | 0
Digital Rectal Exam - Soft Tissue Scarring [Number; unit: participants]
  Yes | 5
  No | 24
Digital Rectal Exam - Hemorrhoids [Number; unit: participants]
  Yes | 2
  No | 27
Digital Rectal Exam - Anal Resting Tone [Number; unit: participants]
  Yes | 27
  No | 2
Endoanal Ultrasound or Magnetic Resonance Imaging Completed [Number; unit: participants]
  Endoanal Ultrasound | 23
  MRI | 6
Endoanal Ultrasound/Magnetic Resonance Imaging - Sphincter Defect [Number; unit: participants]
  Yes | 10
  No | 19
Endoanal Ultrasound/Magnetic Resonance Imaging - Extent of Sphincter Defect [Mean (Standard Deviation); unit: degrees] — Data from 10 subjects who had a sphincter defect. Defects are measured on 0-360 degree scale.
  degrees | 95.0 (50.2)

OUTCOME MEASURES:

1. Primary Outcome: Fecal Incontinence Incidence From Baseline (Pre-treatment) Through 24 Months Post-treatment
Description: Includes solid and liquid stools, as measured by the mean rate obtained using a subject-reported bowel diary. The 3 month post-treatment visit was the primary endpoint time period.
Time Frame: Baseline (pre-treatment), 6 Week, 3 Month, 6 Month, 12 Month and 24 Month post-treatment
Population: The FI Bowel Diary was completed by the number of subjects at each visit as follows:
  Baseline: N=29, 6 Week: N=26, 3 Month: N=27, 6 Month: N=24, 12 Month: N=23, 24 Month: N=26
Measure: Mean (Standard Deviation); unit: Number of FI episodes/14 day period
Arm/Group | TOPAS
Number analyzed (Participants) | 29
Number of FI episodes/14 day period
  Baseline (n = 29) | 6.9 (5.1)
  6 Week (n = 26) | 3.0 (3.2)
  3 Month (primary endpoint time period, n = 27) | 3.7 (4.4)
  6 Month (n = 24) | 3.7 (5.0)
  12 Month (n = 23) | 3.1 (4.1)
  24 Month (n = 26) | 3.5 (3.4)

2. Secondary Outcome: Incidence Rate of Complications During the 24 Month Post-Treatment Follow-up Period
Description: Complications are defined as all adverse events reported during the 24 month follow-up period including serious/non-serious events and events related/not related to the device and/or procedure. Incidence rate is calculated as: (total number of adverse events reported in the 24 month follow-up period) / (total number of subjects implanted = 29)
Time Frame: Through 24 month post-treatment
Population: Includes all subjects implanted with the TOPAS device
Measure: Number; unit: events per 24 months/participant
Arm/Group | TOPAS
Number analyzed (Participants) | 29
events per 24 months/participant
  All Adverse Events | 2.34
  Device and/or Procedure-Related Adverse Events | 0.66
  All Serious Adverse Events | 0.17
  Device and/or Procedure Related Serious Events | 0.03

3. Secondary Outcome: Fecal Incontinence Symptoms as Measured by the Wexner Score
Description: The Wexner Score (also known as the Cleveland Clinic Florida Incontinence Score) is a subject-completed questionnaire that asks about the frequency of incontinence to gas, liquid, solid, of the need to wear pads, and of lifestyle changes (scored on a frequency scale from 0 (=absent) to 4 (daily). An overall Wexner Score is computed from these five components and a score of 0 means perfect control and 20 means complete incontinence.
Time Frame: Baseline (pre-treatment), 6 Week, 3 Month, 6 Month, 12 Month and 24 Month post-treatment
Population: The Wexner Score was completed by the number of subjects at each visit as follows:
  Baseline: N=29, 6 Week: N=29, 3 Month: N=26, 6 Month: N=25, 12 Month: N=25, 24 Month: N=23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 29
units on a scale
  Baseline (n = 29) | 13.2 (2.6)
  6 Week (n = 29) | 7.6 (4.0)
  3 Month (n = 26) | 7.5 (4.1)
  6 Month (n = 25) | 8.5 (4.4)
  12 Month (n = 25) | 8.7 (4.0)
  24 Month (n = 23) | 9.9 (4.4)

4. Secondary Outcome: Fecal Incontinence Symptoms as Measured by Symptom Severity Scale in Fecal Incontinence
Description: The Symptom Severity Scale in Fecal Incontinence is a subject-completed questionnaire that asks about the symptoms of fecal incontinence in the following areas: frequency, stool composition, stool amount, and degree of urgency. The total score is measured on a 0 (best) to 13 (worst) scale. Scores of 1-6, 7-10, and 11-13 were categorized as mild, moderate, and severe fecal incontinence, respectively.
Time Frame: Baseline (pre-treatment), 6 Week, 3 Month, 6 Month, 12 Month and 24 Month post-treatment
Population: The Symptom Severity Scale in Fecal Incontinence was completed by the number of subjects at each visit as follows:
  Baseline: N=29, 6 Week: N=29, 3 Month: N=26, 6 Month: N=25, 12 Month: N=25, 24 Month: N=23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 29
units on a scale
  Baseline (n = 29) | 10.1 (1.4)
  6 Week (n = 29) | 7.4 (2.4)
  3 Month (n = 26) | 7.2 (2.7)
  6 Month (n = 25) | 7.5 (2.8)
  12 Month (n = 25) | 8.0 (2.7)
  24 Month (n = 23) | 8.1 (2.4)

5. Post Hoc Outcome: Percentage of Subjects With Greater Than or Equal to a 50 Percent Reduction in FI Episodes From Baseline
Description: Includes solid and liquid stools, as measured by a subject-reported bowel diary
Time Frame: 6 Weeks, 3 Month, 6 Month, 12 Month and 24 Month post-treatment
Population: Two subjects were enrolled who recorded no FI episodes at baseline and were excluded from this analysis. Missing data was not imputed and was considered a treatment failure.
  The Bowel Diary was completed by the number of subjects at each visit as follows:
  6 Week: N=24, 3 Month: N=25, 6 Month: N=22, 12 Month: N=21, 24 Month: N=24
Measure: Number (90% Confidence Interval); unit: percentage participants
Arm/Group | TOPAS
Number analyzed (Participants) | 27
percentage participants
  6 Week (n = 24) | 59.3 [41.7 to 75.2]
  3 Month (n = 25) | 63.0 [45.3 to 78.3]
  6 Month (n = 22) | 51.9 [34.7 to 68.7]
  12 Month (n = 21) | 40.7 [24.8 to 58.3]
  24 Month (n = 24) | 55.6 [38.2 to 72.0]

6. Secondary Outcome: Quality of Life Assessment as Measured by Fecal Incontinence Quality of Life
Description: The Fecal Incontinence Quality of Life Assessment is a subject-completed questionnaire. It is measured in each of four areas of depression (7 items), lifestyle (10 items), coping (9 items), and embarrassment (3 items). Area scores are measured on a 1 (worse) to 4 (best) scale and are each the average of their component individual item scores measured on the same scale.
Time Frame: Baseline (pre-treatment), 3 Month, 6 Month, 12 Month and 24 Month post-treatment
Population: The Fecal Incontinence Quality of Life Assessment was completed by the number of subjects at each visit as follows:
  Baseline: N=29, 3 Month: N=26, 6 Month: N=25, 12 Month: N=25, 24 Month: N=23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 29
units on a scale
  Depression - Baseline (n = 29) | 2.7 (0.8)
  Depression - 3 Month (n = 26) | 3.3 (0.7)
  Depression - 6 Month (n = 25) | 3.2 (0.8)
  Depression - 12 Month (n = 25) | 3.3 (0.8)
  Depression - 24 Month (n = 23) | 3.3 (0.7)
  Lifestyle - Baseline (n = 29) | 2.7 (0.8)
  Lifestyle - 3 Month (n = 26) | 3.4 (0.7)
  Lifestyle - 6 Month (n = 25) | 3.4 (0.7)
  Lifestyle - 12 Month (n = 25) | 3.3 (0.8)
  Lifestyle - 24 Month (n = 23) | 3.5 (0.7)
  Coping - Baseline (n = 29) | 1.9 (0.5)
  Coping - 3 Month (n = 26) | 2.9 (0.8)
  Coping - 6 Month (n = 25) | 2.8 (0.8)
  Coping - 12 Month (n = 25) | 2.8 (0.9)
  Coping - 24 Month (n = 23) | 2.8 (0.9)
  Embarrassment - Baseline (n = 29) | 1.8 (0.6)
  Embarrassment - 3 Month (n = 26) | 2.9 (0.9)
  Embarrassment - 6 Month (n = 25) | 2.9 (1.0)
  Embarrassment - 12 Month (n = 25) | 3.0 (0.9)
  Embarrassment - 24 Month (n = 23) | 2.9 (1.0)

7. Secondary Outcome: Pain Intensity as Measured by the Pain Intensity Scale
Description: The Pain Intensity Scale is a subject completed questionnaire. Scores are measured on 0 (no pain) to 10 (worst possible pain) scale.
Time Frame: Baseline (pre-treatment), 6 Week post-treatment
Population: The Pain Intensity Scale was completed by the number of subjects at each visit as follows:
  Baseline: N=29, 6 Week: N=29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 29
units on a scale
  Baseline (n = 29) | 1.0 (1.5)
  6 Week (n = 29) | 0.4 (0.8)

8. Secondary Outcome: Intra- and Peri-Surgical Parameters: Length of Procedure
Time Frame: Duration of the device implant procedure
Population: All enrolled/implanted subjects were included in this analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TOPAS
Number analyzed (Participants) | 29
minutes | 23 (8)

9. Secondary Outcome: Intra- and Peri-Surgical Parameters: Length of Hospital Stay
Time Frame: Length of the hospital stay for the device implant procedure
Population: All enrolled/implanted subjects were included in this analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TOPAS
Number analyzed (Participants) | 29
hours | 22.6 (11.6)

10. Secondary Outcome: Intra- and Peri-Surgical Parameters: Estimated Blood Loss During Implant Procedure
Time Frame: Duration of the device implant procedure (an average of 23 minutes)
Population: All enrolled/implanted subjects were included in this analysis
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | TOPAS
Number analyzed (Participants) | 29
ml | 15 (13)

11. Other Pre Specified Outcome: Anal Manometry: Maximum Resting Pressure
Time Frame: Baseline (pre-treatment), 6 Month post-treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TOPAS
Number analyzed (Participants) | 29
mmHg
  Baseline (n = 28) | 29.2 (23.2)
  6 Month (n = 20) | 37.7 (25.8)

12. Other Pre Specified Outcome: Anal Manometry: Maximum Squeeze Pressure
Time Frame: Baseline (pre-treatment), 6 Month post-treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TOPAS
Number analyzed (Participants) | 29
mmHg
  Baseline (n = 28) | 53.2 (38.7)
  6 Month (n = 20) | 51.8 (32.9)

13. Other Pre Specified Outcome: Anal Manometry: Rectal First Sensation
Time Frame: Baseline (pre-treatment), 6 Month post-treatment
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | TOPAS
Number analyzed (Participants) | 29
cc
  Baseline (n = 29) | 37.6 (22.3)
  6 Month (n = 23) | 41.7 (30.0)

14. Other Pre Specified Outcome: Anal Manometry: Maximum Tolerable Volume
Time Frame: Baseline (pre-treatment), 6 Month post-treatment
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | TOPAS
Number analyzed (Participants) | 29
cc
  Baseline (n = 26) | 115.3 (52.4)
  6 Month (n = 20) | 126.3 (49.6)

15. Other Pre Specified Outcome: Pudendal Nerve Terminal Motor Latency
Description: Pudendal Nerve Terminal Motor Latency is a measure of the time it takes for stimulation of the pudendal nerve to elicit contraction of the pelvic floor muscles and anal sphincter. It is a surrogate marker of pudendal nerve injuries and a means of ascertaining whether anal sphincter weakness is attributable to pudendal nerve injury, sphincter defect, or both.
Time Frame: Baseline (pre-treatment), 6 Month post-treatment
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TOPAS
Number analyzed (Participants) | 29
msec
  Baseline - Right Pudendal Nerve Latency (n = 16) | 3.3 (2.6)
  6 Month - Right Pudendal Nerve Latency (n = 10) | 3.8 (2.8)
  Baseline - Left Pudendal Nerve Latency (n = 17) | 2.9 (2.4)
  6 Month - Left Pudendal Nerve Latency (n = 12) | 3.1 (2.3)

ADVERSE EVENTS:
Time Frame: From implant to 24 months post-treatment
Description: The relationship of all AEs to the procedure and/or device was assessed by the investigator. Events were classified as "definitely not", "remotely", "possibly", "probably" or "definitely" related to the procedure/device. All AEs underwent blinded adjudication for coding and serious determination by the Coordinating Investigator
Arm/Group | TOPAS
Serious Adverse Events (participants affected / at risk) | 5/29
Other Adverse Events (participants affected / at risk) | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOPAS (N=29)
Low Back Pain/Disk Herniation (Nervous system disorders) | 1 (1) — Severe low back pain into legs. Admitted into hospital - MRI completed and indicated L2 - L3 disk herniated. Surgery for L2-L3 disk herniation. Related to procedure but not device. Onset = 3 days post implant.
Blood Clot in Lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject states that she had "2 blood clots in her lungs" that caused her to be hospitalized. Not related to device or procedure. Onset = 541 post implant.
Right Leg Cellulitis (Infections and infestations) | 1 (1) — Ruled out deep vein thrombosis. Hospital admit 5/9/09 and discharges 5/13/09. Treated with vancomycin and rocephin. Not related to device/procedure. Onset = 334 days post implant.
Costochondoritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient was admitted to medical center for right wall chest pain. Negative for pulmonary embolism, electrocardiogram = normal sinus rhythm. Not related to device or procedure. Onset = 136 days post implant,
Carpel Tunnel (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient had carpel tunnel requiring surgical release. Not related to device or procedure. Onset = 733 days from implant.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOPAS (N=29)
Urinary Incontinence (De Novo) (Renal and urinary disorders) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4)
Dyspareunia (De Novo) (Reproductive system and breast disorders) | 3 (3)
Worsening Fecal Incontinence (Gastrointestinal disorders) | 3 (3)
Infection (other than urinary tract infection) (Infections and infestations) | 3 (3)
Abnormal Uterine Bleeding (De Novo) (Reproductive system and breast disorders) | 1 (2)
Worsening Vaginal Prolapse (Reproductive system and breast disorders) | 2 (2)
Worsening Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Leg Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Worsening Depression (Psychiatric disorders) | 2 (2)
Erosion (non-TOPAS Mesh Device) (Reproductive system and breast disorders) | 1 (1)
Vaginal Prolapse (De Novo) (Reproductive system and breast disorders) | 1 (1)
Persistent Vaginal Discharge (Reproductive system and breast disorders) | 1 (1)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Excessive Internal Fibrosis (Reproductive system and breast disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (unclassified) (Investigations) | 13 (28)

LIMITATIONS AND CAVEATS:
This study was not powered to statistically evaluate device performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less